CLINICAL TRIAL: NCT04662229
Title: Efficacy of Low Frequency Eco-guided Percutaneous Electric Stimulation on Handgrip Strength: A Single-blinded Pilot Study
Brief Title: Efficacy of Eco-guided PENS on Handgrip Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PENS-Gifto
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-01

CONDITIONS: Electrical Stimulation; Neuromodulation
Keywords: PENS; low-frecuency stimulation; handgrip strength; percutamos electrical stimulation; Neuromodulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: 10 hz stimulatión (Experimental): Eco-guided percutaneous electrical stimulation application of low frequency electrical current at 10 hz, 240 microsecond, over the median and ulnar nerve in the arm, for 1 minute on each nerve. The intensity of the current will reach the excitomotor threshold, causing visible but comfortable contractions.
  Interventions: Device: Eco-guided Percutaneous Electrical Stimulation
- Sham stimulation (Sham Comparator): Application of the needles only on the median and ulnar nerve of the arm, for 1 minute on each nerve without current intensity and a sound will be applied.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Eco-guided Percutaneous Electrical Stimulation — Pointer 10 hz. A symetric, biphasic current of 10 hz and 240 microsecond. The stimulation intensity will be reaching the excitomotor threshold, producing visible but comfortable contractions.
  Arms: Experimental: 10 hz stimulatión
Device: Sham stimulation — Application of the needles only on the median and ulnar nerve of the arm, for 1 minute on each nerve without current intensity and applying a son.
  Arms: Sham stimulation

SUMMARY:
Low-frequency percutaneous electrical stimulation is the application of an electrical current of <1000Hz through acupuncture needles located on the epineurium of the peripheral nervous system.

The hypothesis is that by placing the electrode, needle, closer to the nerve, a greater stimulation of the same will be achieved, thus being able to obtain greater effects. The goal is to determine if this technique has any effect on grip strength in the short term.

DETAILED DESCRIPTION:
Single-blind randomized clinical trial of n = 12 healthy subjects. 4 assessments of the grip strength of the non-dominant hand will be made using a digital dynamometer, by a blinded investigator. A V0-pre-intervention, a V1-post-intervention, a V2 at 24 hours and a V3 at 10 days after the intervention. Subjects will be randomly assigned by EPIDAT 3.1, to an experimental group or a control group, with n = 6 each group. In the experimental group, an ultrasound-guided percutaneous electrical stimulation will be performed. With a pointer, a symmetrical biphasic low-frequency current of 10 Hz and 240 microseconds will be applied to the median nerve and ulnar nerve, until reaching the excitomotor threshold, with applications of 10 seconds and rests of 5 seconds until reaching a stimulation of 1 minute. total over each nerve. In the control group, the same invasive procedure will be performed, but no type of electrical stimulation will be applied.

Statistical analysis will be performed by another blinded assessor, using IBM SPSS Statistics 24. A two-factor ANOVA (intervention-time) with Bonferroni correction will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Ability to perform all clinical tests and understand the study process, as well as obtaining informed consent.
* Tolerance to the application of electrotherapy.
* That they have not diagnosed any pathology.
* They do not present a contraindication to puncture and / or the application of electric currents.

Exclusion Criteria:

* Neuromuscular disease.
* Epilepsy.
* Trauma, surgery or pain affecting the upper limb.
* Osteosynthesis material in the upper limb.
* Diabetes.
* Cancer.
* Cardiovascular disease.
* Pacemaker or other implanted electrical device.
* Take any drug (NSAIDs, corticosteroids, antidepressants, analgesics, antiepileptics, ...) during the study and in the previous 7 days.
* Presence of tattoos or other external agent introduced into the treatment or assessment area.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Hand-grip Strength | baseline at 0 minutes
  Muscle strength will be measured with a dynamometer and will be expressed in Kgs.
Hand-grip Strength | Time Frame: immediately after intervention at 1 minute
  Muscle strength will be measured with a dynamometer and will be expressed in Kgs.
Hand-grip Strength | Time Frame: 24 hours after intervention
  Muscle strength will be measured with a dynamometer and will be expressed in Kgs.
Hand-grip Strength | Time Frame: 10 days after intervention
  Muscle strength will be measured with a dynamometer and will be expressed in Kgs.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Avendaño-Coy, PhD, Study Director — Castilla-La Mancha University
Locations (1):
- Castilla-La Mancha University, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alvarez DM, Serrano-Munoz D, Fernandez-Perez JJ, Moreno JS, Gomez-Soriano J, Avendano-Coy J. The effect on handgrip strength of low-frequency percutaneous electric stimulation applied to the median and cubital nerves: A randomized, double-blind controlled trial. Anat Rec (Hoboken). 2023 Apr;306(4):720-727. doi: 10.1002/ar.24887. Epub 2022 Feb 15. PMID 35166034